CLINICAL TRIAL: NCT06526052
Title: Targeting Negative Affect Through Mindfulness Training in Youth at Risk for Internalizing Problems (R33)
Brief Title: A Randomized Controlled Trial Testing the Effect of the Youth Mindful Awareness Program on Negative Affect (YMAP2).
Acronym: YMAP2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Garber, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R33MH119270 (NIH); 4R33MH119270-03 (NIH)
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Prevention; Control
Keywords: Adolescents; Mindfulness; Internalizing

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three conditions in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will be unaware (masked) of the condition to which participants are randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Program (Experimental): The Mindfulness Program is an online, coached intervention that teaches mindfulness activities such as calm breathing, listening, acceptance, gratitude, and compassion. Participants meet with their coach weekly for nine 30-minute, weekly sessions in which they learn mindfulness skills and practice using the mindfulness exercises between sessions. Meetings are done remotely (e.g., Zoom).
  Interventions: Behavioral: Mindfulness Program
- Supportive Active Comparison (Active Comparator): The Supportive Active condition involves participants meeting remotely (e.g., Zoom) with a coach for nine 30-minute, weekly sessions during which teens discuss their thoughts and feelings about things going on in their life. Coaches are instructed to use active listening, open-ended questions, empathy, reflection, and unconditional positive regard. Between sessions, teens use expressive writing to describe and understand their thoughts and feelings about situations in their life.
  Interventions: Behavioral: Active Comparator
- Control (No Intervention): This is an assessment only control condition. Participants complete all of the same measures as do youth in the other two conditions at the same time points (i.e., baseline, post-intervention (about 10 weeks after baseline) and at a six-month follow-up.

INTERVENTIONS:
Behavioral: Mindfulness Program — Online, coached mindfulness training program
  Arms: Mindfulness Program
Behavioral: Active Comparator — Remote meetings with a supportive coach
  Other Names: Supportive Active Comparison
  Arms: Supportive Active Comparison

SUMMARY:
The goal of this randomized clinical trial is to compare the effects of an online mindfulness program to an active supportive comparison condition and a no-intervention control group on reducing and preventing mood and anxiety symptoms in at-risk youth. Youth who are high on trait negative affect will be randomized to one of the three conditions. The primary outcomes of interest are reductions in momentary negative affect and internalizing problems in adolescents ages 12 to 17 years old. All participants will be evaluated prior to being randomized, after the 9-session intervention period, and at a 6-month follow-up.

The first hypothesis is that the mindfulness intervention will predict decreases in stressor-reactive momentary negative affect and internalizing symptoms. The second hypothesis is that changes in momentary negative affect will partially account for the effects of the mindfulness intervention on internalizing symptoms.

DETAILED DESCRIPTION:
Rates of anxiety and depression in youth are substantial, causing a major unmet need for effective prevention and treatment. A salient risk factor for anxiety and depression is negative affectivity - a partially heritable propensity to experience and express more frequent, intense, and enduring aversive emotional states. Prior longitudinal studies have shown that elevated trait negative affectivity (tNA) during mid-adolescence predicted internalizing disorders later in adolescence and early adulthood, and this relation was partially mediated by changes in momentary negative affect (mNA) measured with ecological momentary assessment (EMA). The conceptual rationale for this investigation is as follows: Trait negative affectivity (tNA) is a risk factor for internalizing symptoms and disorders. tNA also predicts higher levels of momentary negative affect (mNA), measured with EMA, which in turn partially accounts for the prospective association between tNA and symptoms of anxiety and depression. Mindfulness interventions reduce both mNA and internalizing symptoms. Given these empirical relations, this study will test whether in youth with high levels of tNA, an online, coached mindfulness program reduces mNA, as measured with EMA, and whether significantly reducing mNA via a mindfulness intervention then prevents the worsening or onset of internalizing problems.

Mindfulness-based interventions have been found to reduce negative affect and internalizing symptoms in children and adolescents. This study will evaluate changes in mNA as a transdiagnostic target of mindfulness-based training in youth at high risk (i.e., high tNA) for internalizing problems, and the degree to which reductions in such mNA partially account for the effects of mindfulness training on internalizing outcomes in youth. This randomized controlled prevention trial will test the extent to which youth assigned to an online, coached mindfulness program as compared to youth in a supportive attention comparison intervention and a no-intervention control condition will show reduced mNA and its two components -- stressor-independent and stressor-reactive momentary negative affect. The mindfulness training will be implemented through mobile technology (e.g., online program). Investigating the efficacy of an online mode of delivery of mindfulness with support of a coach can advance the prevention of internalizing psychopathology in a manner that could be disseminated broadly. Such technology would improve access to care for youth who can be easily identified as being vulnerable to internalizing problems due to having high levels of tNA.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12, 13, 14, 15, 16, 17
* Parental Consent
* Participant Assent
* Live in Illinois, California, or Tennessee

Exclusion Criteria:

* current diagnosis of an anxiety or depressive disorder with significant clinical impairment
* current alcohol or substance use disorder
* current serious suicidal ideation or behavior
* lifetime diagnosis of bipolar disorder, schizophrenia, autism, conduct disorder, or developmental delay
* reading level below 4th grade
* not English speaking at a level that would allow them to participate in the intervention and assessments

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Assessment of Momentary Negative Affect and Stress | week 10
  EMA involves assessments four times a day for 7 days. The measures of momentray negative affect (mNA) from the EMA are Stressor-Independent (mNA-SI), Stressor-Reactive (mNA-SR), and average mNA.
Internalizing symptoms factor | week 12
  The internalizing symptoms factor is based on a principal components analyses (PCAs) of the change scores for child symptom scales including the Negative Affectivity (NA-15), the Patient Health Question 9 (PHQ9 - measure of depressive symptoms), Generalized Anxiety Disorder 7 (GAD7 - measure of symptoms of anxiety), and the Screen for Child Anxiety Related Disorders (SCARED).

SECONDARY OUTCOMES:
Internalizing symptoms factor | Six-months
  The internalizing symptoms factor is based on a principal components analyses (PCAs) of the change scores for child symptom scales including the Negative Affectivity (NA-15), the Patient Health Question 9 (PHQ9 - measure of depressive symptoms), Generalized Anxiety Disorder 7 (GAD7 - measure of symptoms of anxiety), and the Screen for Child Anxiety Related Disorders (SCARED).
Diagnoses of Anxiety and Depressive Disorders | week 12
  The Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime Version assesses diagnoses at and since baseline and screens for exclusion criteria at baseline (Kaufman et al., 1997).
Diagnoses of Anxiety and Depressive Disorders | Six-months
  The Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime Version (KSADs-PL) assesses diagnoses of anxiety and depressive disorders since the post-intervention assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Megan M Saylor, PhD, Study Chair — Vanderbilt University
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Northwestern University, Evanston, Illinois
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No